CLINICAL TRIAL: NCT02182713
Title: Combivent vs. Salbutamol in Patients With Metacholine Induced Bronchospasm
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1012.36
Record Dates: First submitted 2014-07-03; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol; Ipratropium

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm 1 - CombiventTM followed by Salbutamol (Experimental)
  Interventions: Drug: Salbutamol sulfate/Ipratropium bromide; Drug: Salbutamol
- Arm 2 - Salbutamol followed by CombiventTM (Active Comparator)
  Interventions: Drug: Salbutamol sulfate/Ipratropium bromide; Drug: Salbutamol

INTERVENTIONS:
Drug: Salbutamol sulfate/Ipratropium bromide — Salbutamol sulfate 120 mcg + Ipratropium bromide 20 mcg per puff
  Other Names: CombiventTM
Drug: Salbutamol — Salbutamol 100 mcg per puff
  Other Names: Ventolin®

SUMMARY:
The purpose of this study was to evaluate whether 2 puffs of fixed combination of aerosolized 120 mcg salbutamol sulphate (equivalent to 100 mcg of the base) + 20 mcg ipratropium bromide confers significant additional protection against metacholine induced bronchoconstriction in asthmatic atopic patients when compared to 2 puffs of aerosolized 100 mcg salbutamol alone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with a diagnosis of asthma according to the American Thoracic Society Criteria
* Patients aged 7 to 12 years inclusive
* Patients able to perform spirometry
* Patients with FEV1 (forced expiratory volume in the first second) ≥ 80% of predicted normal value after saline
* Patients with PD20 (provocative dose that reduces FEV1 by 20 %) metacholine lower than 8 mg/ml
* Patients or responsible relatives willing and able to sign an informed consent form

Exclusion Criteria:

* Patients on treatment for or suspected as having glaucoma
* Patients with known allergy of contra-indications to either salbutamol, ipratropium or their excipients
* Patients suspected on clinical grounds to have pneumonia, pneumothorax or pneumomediastinum
* Patients with a history of chest surgery
* Patients with other respiratory conditions if diagnosed. These include pulmonary fibrosis, bronchiectasis, cystic fibrosis, sarcoidosis, pulmonary tuberculosis, pulmonary complications of AIDS
* Patients requiring drugs for the treatment of the acute asthma attack other than the study drugs or oxygen
* Patients who have been previously recruited into this study
* Patients with myocardiopathy, pulmonary edema or other life threatening diseases, which in the judgement of the pediatrician precludes their entry into the study
* Patients with obvious or previously diagnosed serious hepatic or renal disease
* Patients who have been under the following drugs within the specified periods of time prior to determination of Baseline FEV1 or metacholine challenge

  * INHALED:
  * Short acting β2 agonists: 6 hours
  * Long acting β2 agonists: 12 hours
  * Ipratropium bromide: 8 hours
  * DSCG (disodium cromoglicate): 7 days
  * Nedocromil: 7 days
  * ORAL:
  * Short acting β2 agonists: 18 hours
  * Anticholinergics: 7 days
  * Short acting theophylline: 24 hours
  * Long acting theophylline: 72 hours
  * Antihistamines: 7 days
  * Astemizole: 3 months
  * Ketotifen: 3 months
  * INHALED or ORAL: Other investigational drugs: 3 months
  * INHALED or ORAL: Corticosteroids: 30 days

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 1998-05; Primary Completion 1998-09 (Actual)

PRIMARY OUTCOMES:
Increase in PD20 (provocative dose that reduce forced expiratory volume at one second (FEV1) by 20%) | Baseline and 30 minutes after treatment

SECONDARY OUTCOMES:
Change from baseline in systolic and diastolic blood pressure | Baseline, 30 and 60 min after treatment
Change from baseline in heart rate | Baseline, 30 and 60 min after treatment
Change from baseline in respiratory rate | Baseline, 30 and 60 min after treatment
Occurrence of adverse events | up to 8 days
SaO2 (oxygen saturation) during metacholine challenge | continuously after adminstration of study drug